CLINICAL TRIAL: NCT00105664
Title: Collaborative Cardiac Care Project (C3P)
Brief Title: Collaborative Cardiac Care Project
Acronym: C3P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHI 02-062
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-10

CONDITIONS: Myocardial Ischemia; Angina Pectoris; Coronary Disease
Keywords: Outcomes Assessment; Primary Health Care; Group Process
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Collaborative care model; Procedure: Group interventions; Procedure: Facilitated consultation

INTERVENTIONS:
Procedure: Collaborative care model
Procedure: Group interventions
Procedure: Facilitated consultation

SUMMARY:
Data from VA-funded studies and the broader literature indicate that chronic stable angina (CSA) is prevalent, under recognized, under treated and associated with reduced quality of life. There are substantial opportunities for improving care of patients with this debilitating and potentially fatal problem. Because primary care providers manage most patients with CSA, efforts to improve care must necessarily involve the primary care delivery system. C3P is composed of a set of interventions employing a Collaborative Care Team model, which has been shown to be effective in managing other chronic illnesses in the primary care setting.

DETAILED DESCRIPTION:
Objectives of the proposed project are to: 1) ascertain whether a collaborative approach to managing CSA in primary care results in better symptom control and quality of life than routine care; 2) assess whether the practice of providers assigned to the intervention group is more consistent with national clinical practice guidelines than that of control providers; 3) assess satisfaction of both patients and providers with this approach to management; and 4) assess marginal cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Providers:

* Staff (MD, PA, NP) or resident (R1, R2)
* at least 1 participating patient

Patients

* assigned to participating provider
* diagnosis consistent with IHD
* 2 visits in past year
* frequent angina symptoms (SAQ freq. score less than 70)

Exclusion Criteria:

Providers:

- No participating patients

Patients:

* cognitive impairment (inability to complete questionnaires and phone interviews)
* non-participating provider
* life expectancy of less than 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2004-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Symptom control, quality of life and satisfaction at one year; improved practitioner compliance with national clinical practice guidelines over the one-year intervention period

SECONDARY OUTCOMES:
Marginal cost effectiveness during one-year study period

CONTACTS AND LOCATIONS:
Overall Officials: Stephan D. Fihn, MD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Result] Wang L, Porter B, Maynard C, Bryson C, Sun H, Lowy E, McDonell M, Frisbee K, Nielson C, Fihn SD. Predicting risk of hospitalization or death among patients with heart failure in the veterans health administration. Am J Cardiol. 2012 Nov 1;110(9):1342-9. doi: 10.1016/j.amjcard.2012.06.038. Epub 2012 Jul 21. PMID 22819429
- [Result] Fihn SD, Bucher JB, McDonell M, Diehr P, Rumsfeld JS, Doak M, Dougherty C, Gerrity M, Heidenreich P, Larsen G, Lee PI, Lucas L, McBryde C, Nelson K, Plomondon ME, Stadius M, Bryson C. Collaborative care intervention for stable ischemic heart disease. Arch Intern Med. 2011 Sep 12;171(16):1471-9. doi: 10.1001/archinternmed.2011.372. PMID 21911632
- [Result] Fan VS, Bridevaux PO, McDonell MB, Fihn SD, Besser LM, Au DH. Regional variation in health status among chronic obstructive pulmonary disease patients. Respiration. 2011;81(1):9-17. doi: 10.1159/000320115. Epub 2010 Aug 17. PMID 20720400